CLINICAL TRIAL: NCT00338442
Title: Safety and Efficacy of Varicella Zoster Immune Globulin (Human) VariZIG in Patients at Risk of Varicella Infection
Status: Approved for marketing | Type: Expanded Access
Sponsor: Cangene Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: VZ-009
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Varicella
Keywords: Immune compromised; Varicella Zoster Virus ( VZV) Infection; Pediatric
MeSH Terms: conditions — Chickenpox; Infections | interventions — varicella-zoster immune globulin

INTERVENTIONS:
Drug: VariZIG™ — Biological / Vaccine

SUMMARY:
This study is to assess VariZIG™ for the treatment of patients at risk for developing serious complications from chicken pox.

DETAILED DESCRIPTION:
In most individuals, chicken pox or varicella zoster (VZV) infections are benign; however, in certain at-risk populations such as immunocompromised patients or infants VZV disease can produce significant morbidity and mortality. In such patients, varicella zoster immune globulin (VZIG) has been used to prevent or reduce the severity of VZV infections in at-risk patients exposed to individuals with active infections. Massachusetts Public Health Biologic Laboratories (Boston, MA) has discontinued manufacture of the only FDA approved VZIG product. Cangene Corporation (Winnipeg, Canada) is conducting this expanded access IND protocol for VariZIG™, which is a purified human immune globulin preparation made from plasma of donors with high anti-varicella antibody titers.

This study is an open label, non-randomized, expanded access study that will make VariZIG™ available to eligible patients for whom there is no alternative licensed treatment while a pivotal study is conducted. The study will begin recruiting in February 2006 and will collect safety and basic efficacy data over 42 days following VariZIG™ administration. Physicians will be required to assess measures of varicella infection as well as provide study specific documentation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Cangene Corporation VariZIG™ release requirement.
* Any of the following at-risk patients exposed to varicella within the previous 96 hours:

  * Immunocompromised pediatric or adult patients.
  * Neonates (less than 1 year of age) and pre-term infants.
  * Pregnant women.
  * Newborns whose mothers had VZV infection shortly before delivery (< 5 days) or after (< 2 days) delivery.
  * Healthy non-immune adults

Exclusion Criteria:

* Hypersensitivity to blood or blood products, including intravenous (IV) or intramuscular (IM) human immunoglobulin preparations.
* Selective immunoglobulin A (IgA) deficiency.
* Evidence of VZV infection.
* Evidence of zoster infection.
* Known immunity to VZV(previous varicella infection or varicella vaccination)
* Severely thrombocytopenic ( platelets < 50 x 10x9 / L )

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-02; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gale, MD, Principal Investigator — FFF Enterprises

REFERENCES:
- [Derived] Gans H, Chemaly RF. Varicella zoster immune globulin (human) (VARIZIG) in immunocompromised patients: a subgroup analysis for safety and outcomes from a large, expanded-access program. BMC Infect Dis. 2021 Jan 11;21(1):46. doi: 10.1186/s12879-020-05656-6. PMID 33430796
- [Derived] Duchon JM, Levin MJ, Gershon AA. Safety and Varicella Outcomes in In Utero-Exposed Newborns and Preterm Infants Treated With Varicella Zoster Immune Globulin (VARIZIG): A Subgroup Analysis of an Expanded-Access Program. J Pediatric Infect Dis Soc. 2020 Sep 17;9(4):449-453. doi: 10.1093/jpids/piz070. PMID 31774916